CLINICAL TRIAL: NCT04843592
Title: Effectiveness of Using SOKARY Mobile Application on Compliance of Patient With Type II Diabetes: A Quasi- Experimental Study
Brief Title: SOKARY Mobile Application With Type II Diabetes
Acronym: DM
Status: Completed | Type: Observational
Sponsor: Magda Bayoumi (Other)
Responsible Party: Sponsor-Investigator, Magda Bayoumi, Lecturer, Beni-Suef University
Organization: Beni-Suef University (Other)
Other Study IDs: EC10082019
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2019-08

CONDITIONS: Type II Diabetes
Keywords: Mobile phone application; DM type II; EGYPT; Compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type II diabetes: using mobile app
  Interventions: Device: SOKARY Mobile

INTERVENTIONS:
Device: SOKARY Mobile — Effectiveness of using SOKARY Mobile Application on compliance of patient with Type II diabetes

SUMMARY:
Android mobile application named (SOKARY)

DETAILED DESCRIPTION:
Android mobile application named (SOKARY) which means diabetes was selected as an example of mobile health application as it has the advantage of Arabic interface, free use it allows users to record his/their blood glucose level, nutrition and physical activity, then provide the user with statistics for those readings. The application also sends notifications to the users such as medication reminders and healthy lifestyle advice.

ELIGIBILITY:
Inclusion Criteria:

* Be familiar with the use of mobile health applications.
* Own a smartphone with an android operating system.
* Able to use the internet either through Wi-Fi network and\or mobile data.

Exclusion Criteria:

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient with type II DM
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
the patient's compliance after using SOKARY mobile app | 3 months
  Increase level of Patients' compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided